CLINICAL TRIAL: NCT07140991
Title: The Effect of Perioperative Hyperglycemia on Anastomotic Leaks in Patients Undergoing Total Gastrectomy: A Retrospective Cohort Study
Brief Title: The Effect of Perioperative Hyperglycemia on Anastomotic Leaks After Total Gastrectomy
Status: Completed | Type: Observational
Sponsor: Taner Abdullah (Other)
Responsible Party: Sponsor-Investigator, Taner Abdullah, MD, Istanbul Saglik Bilimleri University
Organization: Istanbul Saglik Bilimleri University (Other)
Other Study IDs: 2025-183
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hyperglycaemia; Total Gastrectomy; Anastomotic Leaks
Keywords: hyperglycaemia; total gastrectomy; anastomotic leak
MeSH Terms: conditions — Hyperglycemia; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hyperglycemia: Patients identified as hyperglycemic in the perioperative period

SUMMARY:
Esophagojejunostomy anastomosis is used in total gastrectomy surgeries. Anastomotic leakage is a serious complication seen after these surgeries and is associated with increased morbidity and mortality. Patients with older age and comorbidities have a higher risk of death following anastomotic leakage.

Perioperative hyperglycemia is frequently observed in patients undergoing major abdominal surgery as a stress response to surgical trauma, leading to surgical complications through mechanisms such as glycogenolysis, lipolysis, gluconeogenesis, decreased insulin sensitivity, and increased insulin resistance. Hyperglycemia is known to increase the risk of postoperative infection, prolong hospital stay, and increase mortality. Additionally, recent studies have shown that it also increases the risk of anastomotic leakage.

DETAILED DESCRIPTION:
Although diabetes mellitus is a known risk factor for anastomotic leaks, there are few studies on the relationship between perioperative hyperglycemia and anastomotic leaks. The primary objective of our study was to demonstrate the relationship between hyperglycemia detected during anastomosis formation in the perioperative period and postoperative anastomotic leaks.

ELIGIBILITY:
Inclusion Criteria:

* elective total gastrectomy
* anastomotic leak after surgery
* age 18-75

Exclusion Criteria:

* emergency procedure
* <18 years
* >75 years
* ASA score > 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was planned as a single-center retrospective study involving patients between the ages of 18 and 75 who underwent total gastrectomy and esophago-jejunostomy anastomosis for benign or malignant reasons.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
postoperative anastomotic leakage | 30 days after surgery
  Patients who developed anastomotic leak after total gastrectomy

SECONDARY OUTCOMES:
diabetic hyperglysemia | intraoperative
  Patients with diabetes but unregulated blood sugar
non-diabetic hyperglysemia | intraoperative
  Patients without diabetes who became hyperglycemic due to surgical stress

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Çağrı Temel, MD, Principal Investigator — Basaksehir Cam ve Sakura State Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No